CLINICAL TRIAL: NCT00048945
Title: Efficacy and Safety Study of Pegasys in the Treatment of Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Purpose: Treatment
Other Study IDs: WV16240
Record Dates: First submitted 2002-11-12; First posted 2002-11-14 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

INTERVENTIONS:
Drug: PEGASYS

SUMMARY:
The purpose of this study is to determine the safety and efficacy of Pegasys + placebo + lamivudine versus lamivudine alone in patients with lamivudine versus lamivudine alone in patients with hepatitis B antigen CHB.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hepatitis B
* Not pregnant

Exclusion Criteria:

* Treatment for hepatitis B in past 6 months
* Other hepatitis infections
* Severe liver disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2002-01 (Actual); Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (57):
- United States (15):
  - Scottsdale, Arizona
  - Downey, California
  - Los Angeles, California
  - Pasadena, California
  - San Francisco, California
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Minneapolis, Minnesota
  - Lincoln, Nebraska
  - Chapel Hill, North Carolina
  - Cedar Creek, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- Australia (2):
  - Concord
  - Herston
- Brazil (4):
  - Campinas
  - Porto Alegre
  - Salvador
  - São Paulo
- Canada (2):
  - Calgary, Alberta
  - Toronto, Ontario
- China (7):
  - Beijing
  - Chengdu
  - Chongqing
  - Guangzhou
  - Hangzhou
  - Hong Kong
  - Shanghai
- France (2):
  - Clichy
  - Lyon
- Germany (6):
  - Berlin
  - Bochum
  - Cologne
  - Düsseldorf
  - Hanover
  - München
- Israel (3):
  - Haifa
  - Petah Tikva
  - Tel Aviv
- Otahuhu, New Zealand
- Poland (3):
  - Bialystok
  - Bydgoszcz
  - Warsaw
- Santurce, Puerto Rico
- Singapore, Singapore
- Seoul, South Korea
- Basel, Switzerland
- Taiwan (4):
  - Kaohsiung City
  - Kwei Shan
  - Tainan
  - Taipei
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Songkhla
- Nottingham, United Kingdom